CLINICAL TRIAL: NCT03723447
Title: A Prospective Randomized Trial of Transversus Abdominis Plane (TAP) INtraoperative Block With Bupivacaine/Dexamethasone aGainst Liposomal Bupivacaine (Exparel®): the TINGLE Trial
Brief Title: Intraoperative TAP Block With Bupivacaine/Dexamethasone Against Liposomal Bupivacaine (Exparel®)
Acronym: TINGLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Karen Zaghiyan, Surgeon Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00053363
Record Dates: First submitted 2018-10-26; First posted 2018-10-29 (Actual); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Pain, Postoperative; Crohn Disease; Inflammatory Bowel Diseases; Colorectal Cancer; Gastrointestinal Cancer; Gastrointestinal Disease; Digestive System Disease; Pain; Pain, Neuropathic; Intestinal Disease
Keywords: transversus abdominis plane block; tap block; liposomal bupivacaine; exparel; dexamethasone; colorectal surgery; regional anesthesia; bupivacaine; surgery; postoperative pain; pain
MeSH Terms: conditions — Pain, Postoperative; Crohn Disease; Inflammatory Bowel Diseases; Colorectal Neoplasms; Gastrointestinal Neoplasms; Gastrointestinal Diseases; Digestive System Diseases; Pain; Neuralgia; Intestinal Diseases | interventions — Bupivacaine; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine/epinephrine/dexamethasone TAP block (Active Comparator): For the bupivacaine/epinephrine/dexamethasone treatment arm, a standard weight-based dose of bupivacaine and epinephrine combined with 8mg dexamethasone will be administered.
  Interventions: Drug: Bupivacaine/epinephrine/dexamethasone
- Liposomal bupivacaine TAP block (Active Comparator): For the liposomal bupivacaine treatment arm, 266mg liposomal bupivacaine (Exparel) will be administered.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Liposomal bupivacaine will be given during the bilateral laparoscopic-guided TAP block given to each patient intraoperatively.
  Other Names: Exparel
  Arms: Liposomal bupivacaine TAP block
Drug: Bupivacaine/epinephrine/dexamethasone — Bupivacaine/epinephrine/dexamethasone will be given during the bilateral laparoscopic-guided TAP block administered to each patient intraoperatively.
  Other Names: Decadron
  Arms: Bupivacaine/epinephrine/dexamethasone TAP block

SUMMARY:
Traditionally, opioids are heavily utilized in treating postoperative pain but they are associated with numerous side effects. The use of the transversus abdominis plane (TAP) blocks have become standard practice to extend the post-operative analgesic window and limit opioid use. A new liposomal-depo formulation of bupivacaine (Exparel) has gained popularity as a long-lasting TAP block medication, but has not been studied in a well-powered clinical trial specifically in colorectal patients nor compared to a bupivacaine/steroid mixture which may offer similar effects. We conduct a prospective randomized prospective randomized study of patients undergoing major laparoscopic colorectal surgery to compare the analgesic effects of a bupivacaine/steroid mixture versus liposomal bupivacaine.

DETAILED DESCRIPTION:
Postoperative pain can pose significant challenges in the postoperative recovery of patients undergoing major colorectal surgery. Traditionally, opioids have played an important role in treating postoperative pain. It is well established that opioids are highly effective in relieving pain; however, opioids are associated with numerous side effects that include nausea, vomiting, constipation, ileus, bladder dysfunction, respiratory depression, pruritus, drowsiness, sedation, and allergic reaction. These opioid side effects, which range in severity, can significantly interfere with discharge home, particularly following colorectal surgery. Significant interest has grown for the use of guided regional anesthesia, specifically the use of the transversus abdominis plane (TAP) block to extend the post-operative analgesic window and ultimately limit opioid use. While bupivacaine formulations including a steroid has been shown to prolong the anesthetic effects of the regional field block, a new liposomal-depo formulation of bupivacaine (Exparel) has gained popularity and has additionally been shown to provide extended analgesia. Although promising data exists surrounding each modality, liposomal bupivacaine has not been studied in a well-powered clinical trial specifically in colorectal patients nor compared to a bupivacaine/steroid mixture.

We are proposing a prospective randomized study of patients undergoing major laparoscopic colorectal surgery to compare the analgesic effects of a bupivacaine/steroid mixture versus liposomal bupivacaine (Exparel). We hypothesize that the liposomal formulation of bupivacaine will provide superior perioperative pain control at 48 hours post-operation measured by total consumed oral morphine equivalents. In addition, we will measure postoperative pain scores, time until ambulation, antiemetic use, length of postoperative hospital stay, postoperative ileus, and adverse events directly related or unrelated to TAP block in the 30-day postoperative period between the three groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Undergoing major laparoscopic colorectal procedure
3. Willingness and ability to sign an informed consent document
4. No allergies to anesthetic or analgesic medications
5. ASA physical status Class I - III
6. Aged 18-90 years

Exclusion Criteria:

1. Refusal to participate in the study
2. Age <18 or > 90 years
3. Pregnancy
4. Contraindications to regional anesthetic including but not limited to:

   1. Patient refusal to regional field blockade
   2. Allergy
   3. Infection at the site of needle insertion
   4. Systemic infection
   5. Bleeding diathesis or coagulopathy (as diagnosed by history or laboratory evaluation)
   6. Liver or renal disease (SCr > 1.5)
5. Chronic opioid use

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zaghiyan, MD, Principal Investigator — Cedars Sinai
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mujukian A, Truong A, Tran H, Shane R, Fleshner P, Zaghiyan K. A Standardized Multimodal Analgesia Protocol Reduces Perioperative Opioid Use in Minimally Invasive Colorectal Surgery. J Gastrointest Surg. 2020 Oct;24(10):2286-2294. doi: 10.1007/s11605-019-04385-9. Epub 2019 Sep 12. PMID 31515761
- [Background] Truong A, Mujukian A, Fleshner P, Zaghiyan K. No Pain, More Gain: Reduced Postoperative Opioid Consumption with a Standardized Opioid-Sparing Multimodal Analgesia Protocol in Opioid-Tolerant Patients Undergoing Colorectal Surgery. Am Surg. 2019 Oct 1;85(10):1155-1158. PMID 31657314
- [Background] Knudson RA, Dunlavy PW, Franko J, Raman SR, Kraemer SR. Effectiveness of Liposomal Bupivacaine in Colorectal Surgery: A Pragmatic Nonsponsored Prospective Randomized Double Blinded Trial in a Community Hospital. Dis Colon Rectum. 2016 Sep;59(9):862-9. doi: 10.1097/DCR.0000000000000648. PMID 27505115
- [Derived] Truong A, Fleshner PR, Mirocha JM, Tran HP, Shane R, Zaghiyan KN. A Prospective Randomized Trial of Surgeon-Administered Intraoperative Transversus Abdominis Plane Block With Bupivacaine Against Liposomal Bupivacaine: The TINGLE Trial. Dis Colon Rectum. 2021 Jul 1;64(7):888-898. doi: 10.1097/DCR.0000000000002008. PMID 34086002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was noted to have chronic opioid use discovered after randomization. They were subsequently excluded from analysis
Period: Overall Study
Arm/Group | Bupivacaine/Epinephrine/Dexamethasone TAP Block | Liposomal Bupivacaine TAP Block
Started | 50 | 51
Completed | 50 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine/Epinephrine/Dexamethasone TAP Block | Liposomal Bupivacaine TAP Block | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [29 to 67] | 42 [29 to 57] | 42 [29 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 22 | 51
  Male | 21 | 29 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 31 | 32 | 63
  Unknown or Not Reported | 14 | 18 | 32
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Cumulative 48-hour Post Surgical Opiate Use (Oral Morphine Equivalent)
Time Frame: 48-hours
Measure: Median (Inter-Quartile Range); unit: Oral morphine equivalents
Arm/Group | Bupivacaine/Epinephrine/Dexamethasone TAP Block | Liposomal Bupivacaine TAP Block
Number analyzed (Participants) | 50 | 51
Oral morphine equivalents | 47 [18 to 112] | 69 [20 to 110]

2. Secondary Outcome: Post-op Pain Score (Visual Analog Scale)
Description: Visual pain scale recordings will be totaled and averaged during the first 72-hours post-surgery. Visual analog scale is determined by nursing staff when assessing pain scores. Scores range from 0-10 with 10 being the most pain. These values are typically interpreted by nursing staff as mild, moderate, or severe pain and pain medication is given accordingly.
Time Frame: 72-hours post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine/Epinephrine/Dexamethasone TAP Block | Liposomal Bupivacaine TAP Block
Number analyzed (Participants) | 50 | 51
score on a scale | 4 [2 to 5] | 4 [2 to 5]

3. Secondary Outcome: Bowel Motility
Description: Time till first bowel movement
Time Frame: 72 hours post-surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Bupivacaine/Epinephrine/Dexamethasone TAP Block | Liposomal Bupivacaine TAP Block
Number analyzed (Participants) | 50 | 51
days | 1 [1 to 2] | 1 [1 to 2]

4. Secondary Outcome: Postoperative Length of Stay
Description: Time from operation until hospital discharge
Time Frame: 30 days post-surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Bupivacaine/Epinephrine/Dexamethasone TAP Block | Liposomal Bupivacaine TAP Block
Number analyzed (Participants) | 50 | 51
days | 3 [2 to 4] | 3 [2 to 5]

5. Secondary Outcome: Postoperative Complications
Description: Medical or surgical complications measured by Clavien-Dindo classification
  Clavien-Dindo grade I: any deviation from normal postoperative course
  * no pharmacological or surgical treatment, endoscopic, or radiological interventions were required. Acceptable therapeutic regiments are drugs such as anti-emetics, antipyretics, analgesics, diuretics, and electrolytes. Wound infections or small abscess requiring incision at bedside is within this category
  Clavien-Dindo grade II: Normal course altered
  * Pharacological management other than in grade 1. Blood transfusions and total parenteral nutrition are also included.
  Clavien-Dindo grade III: complications that require intervention of various degrees
  * management of these complications require an intervention under local anesthesia or general or epidural anesthesia
  Clavien-Dindo grade IV: complications threatening the life of a patient
  * manifesting in organ dysfunction, including dialysis
Time Frame: 30 days post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine/Epinephrine/Dexamethasone TAP Block | Liposomal Bupivacaine TAP Block
Number analyzed (Participants) | 50 | 51
Participants
  None | 29 | 32
  Clavien-Dindo grade I | 7 | 2
  Clavien-Dindo grade II | 8 | 7
  Clavien-Dindo grade III | 6 | 10

ADVERSE EVENTS:
Time Frame: Data was collected for each patient for a maximum period of 3 months postoperatively.
Description: Adverse events are defined by complications or unexpected sequelae as a result of TAP block administration
Arm/Group | Bupivacaine/Epinephrine/Dexamethasone TAP Block | Liposomal Bupivacaine TAP Block
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 0/50 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT03723447/Prot_SAP_000.pdf